CLINICAL TRIAL: NCT07067606
Title: Role of Musculoskeletal Ultrasound for Early Detection of Synovitis in SLE Patient and Its Correlation With Disease Activity and Neutrophil-to-C3 Ratio.
Status: Not yet recruiting | Type: Observational
Sponsor: Mervat Sayed Kamal Sayed (Other)
Responsible Party: Sponsor-Investigator, Mervat Sayed Kamal Sayed, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: musculoskeletal US SLE
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Musckloskeletal US
Keywords: muskluskeletal US - SLE

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound contrast — All participants will be subjected to full history taking, full clinical examination, laboratory investigations (complete blood count, erythrocyte sedimentation rate [ESR], C-reactive protein [CRP], blood urea, serum creatinine, serum glutamic-oxaloacetic transaminase [SGOT], serum glutamate-pyruvate transaminase [SGPT], immunological tests (antinuclear and anti-DNA antibodies and C3 and C4 levels), urine analysis, and 24-h urinary protein). SLE disease activity index (SELDAI) will be also calculated for every patient. (8) Musculoskeletal examination with power Doppler, the ultrasound examination will be performed at the musculoskeletal ultrasonography unit at the rheumatology division of the internal medicine department. Bilateral musculoskeletal US examinations of hands and wrists with power Doppler (PD) evaluation will be done for all patients. US examinations were performed using the standardized scanning technique according to EULAR guidelines for musculoskeletal US in rheumatolog

SUMMARY:
Systemic lupus erythematosus (SLE) is a clinically common autoimmune disease characterized by abnormal immune response to autologous tissue, eventually resulting in systemic disorders and diverse clinical manifestations. The prevalence of women is significantly higher than that of men.

Musculoskeletal and joint affection represents one of the most common manifestations of systemic lupus erythematosus (SLE), and 95% of them have either arthralgia or arthritis during their disease course.

SLE arthropathy has main three different clinical types: nondeforming nonerosive arthritis; the most common type, deforming nonerosive arthropathy (Jaccoud's arthropathy) which has no bone erosions on conventional radiography and exists in up to 15% of the patients and erosive arthropathy (rhupus syndrome) which is overlap syndrome between rheumatoid arthritis (RA) and SLE and exist in <5% of lupus patients.

In clinical practice, most lupus patients who have joint and tendon pains often have no apparent inflammation during physical examination. Joint and tendon inflammation has been documented in musculoskeletal ultrasound in patients without any signs of arthritis, thus suggesting the role of ultrasound in the evaluation of patients with nonspecific musculoskeletal manifestations such as arthralgia. And detection of the presence of underlying subclinical inflammatory changes.

Components of lymphocytes, antibodies, inflammatory cytokines, and complements in peripheral circulation vary among different active stages of SLE. Patients with higher disease activity often damage tissues and organs, many of which even threaten life. It is of great significance in SLE management to early and accurately determine the disease activity of patients.

We will investigate the role of musculoskeletal ultrasound for early detection of synovitis in SLE patients and its correlation with disease activity and neutrophil-to-C3 ratio (NC3R).

DETAILED DESCRIPTION:
All participants will be subjected to full history taking, full clinical examination, laboratory investigations (complete blood count, erythrocyte sedimentation rate [ESR], C-reactive protein [CRP], blood urea, serum creatinine, serum glutamic-oxaloacetic transaminase [SGOT], serum glutamate-pyruvate transaminase [SGPT], immunological tests (antinuclear and anti-DNA antibodies and C3 and C4 levels), urine analysis, and 24-h urinary protein). SLE disease activity index (SELDAI) will be calculated for every patient.

Musculoskeletal examination with power Doppler, the ultrasound examination will be performed at the musculoskeletal ultrasonography unit at the rheumatology division of the internal medicine department. Bilateral musculoskeletal US examinations of hands and wrists with power Doppler (PD) evaluation will be done for all patients. US examinations were performed using the standardized scanning technique according to EULAR guidelines for musculoskeletal US in rheumatology.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients without musculoskeletal manifestations diagnosed according to European League against Rheumatism (EULAR) and the American college of Rheumatology (ACR)criteria for classification of SLE.

Exclusion Criteria:

* • Overlap syndrome as rhupus patients, those with trauma, osteoarthritis, surgery of hand and wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: non probability
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Role of musculoskeletal ultrasound for early detection of synovitis in SLE patient and its correlation with disease activity and neutrophil-to-C3 ratio. | baseline
  early detection of synovitis in SLE patient

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus. Arthritis Rheumatol. 2019 Sep;71(9):1400-1412. doi: 10.1002/art.40930. Epub 2019 Aug 6. PMID 31385462